CLINICAL TRIAL: NCT01802203
Title: trūFreeze® Spray Cryotherapy Patient Registry
Status: Completed | Type: Observational
Sponsor: US Endoscopy Group Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Barrett Esophagus; Esophageal Dysplasia; Esophageal Neoplasm; Esophageal Stenosis; Bronchial Neoplasm; Stenosis of Bronchus or Trachea
Keywords: Barrett esophagus; Esophageal dysplasia; Upper gastrointestinal squamous dysplasia; Esophageal cancer; Endobronchial cancer; Central airway cancer; Central airway precancerous disease; Central airway granulation tissue; Central airway papillomatosis; Central airway sarcoidosis; Central airway tuberculosis; Tracheal stenosis; Bronchial stenosis
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Esophageal Stenosis; Bronchial Neoplasms; Tracheal Diseases; Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- truFreeze spray cryotherapy: truFreeze Spray Cryotherapy administered as routine clinical care
  Interventions: Device: truFreeze Spray Cryotherapy

INTERVENTIONS:
Device: truFreeze Spray Cryotherapy — spray cryotherapy

SUMMARY:
To collect efficacy and outcomes data related to the use of trūFreeze® spray cryotherapy for the treatment of unwanted tissue in the pulmonary and gastrointestinal settings.

DETAILED DESCRIPTION:
This is a prospective, multi-center registry of patients who are currently undergoing spray cryotherapy using the trūFreeze® device. The registry population consists of patients who are being treated using the spray cryotherapy trūFreeze® device for the removal of unwanted tissue, such as malignant or pre-malignant conditions in the pulmonary or gastrointestinal settings.

Patients eligible to participate in the registry will have disease and treatment specific data collected throughout therapy and long-term follow-up. Subjects will be considered to have completed the registry when data from the 5 year follow-up visit has been collected. The beginning of the follow-up period commences with the first endoscopic treatment session.

Subjects may be withdrawn prior to this for any of the following reasons:

1. Death, or
2. Lost to Follow-Up, or
3. Withdrawal of consent, or
4. Discontinuation by the investigator. Three attempts at contact using two different methods are required prior to determination that the subject is lost to follow-up. Attempts at contact must be with certified letters OR documented telephone contact.

The registry will utilize electronic case report forms using a web-based platform housed at the University of North Carolina at Chapel Hill. Access to the database will be limited to individuals involved in the research registry and will require a unique user ID and password. All access to the database and web-based application will be encrypted (HTTPS) and electronic systems compliant with applicable privacy and security regulations. To maintain patient confidentiality, all subjects will be assigned a registry identification number, and this will be the only link between subject identity and treatment information. Read-only access will be provided to any personnel who is not an administrator or responsible for data entry.

All data requested on the case report form must be recorded. All missing data must be explained. The system allows sites to directly enter data electronically, however sites are still responsible for ensuring they have source documents that support all data entered electronically that are separate and verifiable. The registry system will maintain an audit trail that captures when electronic entries are changed, what the change was, and who made the change.

The investigators will ensure the capability for inspections of applicable registry-related facilities (e.g. pharmacy, diagnostic laboratory, etc.). The registry will be monitored by the sponsor, and allow auditing by the Institutional Review Board, government regulatory bodies, and University compliance and quality assurance groups of all registry related documents (e.g. source documents, regulatory documents, data collection instruments, registry data, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. GI conditions include:

   * Barrett's Esophagus (BE) with or without dysplasia
   * Squamous dysplasia
   * Esophageal cancer, any stage
2. Pulmonary conditions include:

   * Any endobronchial cancerous or precancerous disease located within the central airways
   * Any non-malignant endobronchial process of the central airways that results in abnormal mucosa (i.e. granulation tissue, papillomatosis, sarcoidosis, tuberculosis, etc.)
   * Tracheal or bronchial stenosis (malignant or benign)
   * Any pleural disease, malignant or benign All subjects are required to be able to provide written informed consent

Exclusion Criteria:

1. Gastrointestinal Exclusion Criteria

   * Contraindication to spray cryotherapy.
   * Prior treatment with spray cryotherapy. Previous or concurrent treatment using other mucosal therapies such as endoscopic mucosal resection or radiofrequency ablation is acceptable.
   * Below 18 years of age
2. Pulmonary Exclusion Criteria

   * Contraindication to spray cryotherapy.
   * Prior treatment with spray cryotherapy. Previous or concurrent treatment using other mucosal therapies is acceptable.
   * Tracheoesophageal fistula.
   * Bronchopleural fistula.
   * Current untreated pneumothorax.
   * Clinically significant hypoxia refractory to supplemental oxygen therapy.
   * Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being treated using the trūFreeze® spray cryotherapy device for the removal of unwanted tissue, such as malignant or pre-malignant conditions in the pulmonary or gastrointestinal (GI) setting.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2013-04; Primary Completion 2022-01 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Collect efficacy and outcome data related to the use of trūFreeze® spray cryotherapy for treatment of unwanted tissue in the pulmonary and gastrointestinal settings. | 5 years
  The registry population consists of patients who are being treated using the trūFreeze® spray cryotherapy device for the removal of unwanted tissue, such as malignant or pre-malignant conditions in the pulmonary or gastrointestinal settings.

SECONDARY OUTCOMES:
Collect safety data related to the use of trūFreeze® spray cryotherapy for treatment in the pulmonary and gastrointestinal settings. | 5 years
  All adverse events occurring during the registry period must be recorded. The clinical course of each event should be followed until resolution, stabilization, or until it has been determined that the registry treatment or participation is not the cause. Serious adverse events that are still ongoing at the end of the Spray Cryotherapy Patient Registry registry period must be followed up to determine the final outcome. Any serious adverse event that occurs after the registry period and is considered to be possibly related to the trūFreeze® spray cryotherapy device or registry participation should be recorded and reported immediately.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, Principal Investigator — University of North Carolina, Chapel Hill; Robert F Browning, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (16):
- United States (16):
  - Scripps Green Hosptial, La Jolla, California
  - University of Colorado Denver, Denver, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - Ochsner Medical Center, Kenner, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - ProHEALTH Care Associates, Lake Success, New York
  - NYU, New York, New York
  - University of Rochester/Strong Memorial Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ahuja Medical Center-CWR University Hosptials, Beachwood, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Heier SK. Evaluation of candidate therapies for ablation of Barrett's in a canine model. Gastrointestinal endoscopy. 1996;43(4):337
- [Background] Pasricha PJ, Hill S, Wadwa KS, Gislason GT, Okolo PI 3rd, Magee CA, Canto MI, Kuo WH, Baust JG, Kalloo AN. Endoscopic cryotherapy: experimental results and first clinical use. Gastrointest Endosc. 1999 May;49(5):627-31. doi: 10.1016/s0016-5107(99)70393-7. PMID 10228263
- [Background] Greenwald BD, Dumot JA, Horwhat JD, Lightdale CJ, Abrams JA. Safety, tolerability, and efficacy of endoscopic low-pressure liquid nitrogen spray cryotherapy in the esophagus. Dis Esophagus. 2010 Jan;23(1):13-9. doi: 10.1111/j.1442-2050.2009.00991.x. Epub 2009 Jun 9. PMID 19515183
- [Background] Grana L, Ablin RJ, Goldman S, Milhouse E Jr. Freezing of the esophagus: histological changes and immunological response. Int Surg. 1981 Oct-Dec;66(4):295-301. PMID 7345039
- [Background] Loprinzi CL, Foote RL, Michalak J. Alleviation of cytotoxic therapy-induced normal tissue damage. Semin Oncol. 1995 Apr;22(2 Suppl 3):95-7. PMID 7740323
- [Background] Rodgers BM, Pappelis P. Profound endoesophageal cryotherapy. Cryobiology. 1985 Feb;22(1):86-92. doi: 10.1016/0011-2240(85)90011-2. PMID 3979079
- [Background] Laugier P, Berger G. Assessment of echography as a monitoring technique for cryosurgery. Ultrason Imaging. 1993 Jan;15(1):14-24. doi: 10.1177/016173469301500102. PMID 8328116
- [Background] Reiser M, Drukier AK, Ultsch B, Feuerbach S. The use of CT in monitoring cryosurgery. Eur J Radiol. 1983 May;3(2):123-8. PMID 6873073
- [Background] Myers B, Donovan W. Cryosurgery of the anus. South Med J. 1977 Jan;70(1):17-8. doi: 10.1097/00007611-197701000-00008. PMID 841369
- [Background] McKelvie P. Cryotherapy in the upper air and food passages. Proc R Soc Med. 1975 Oct;68(10):610. doi: 10.1177/003591577506801005. No abstract available. PMID 54925
- [Background] Kuflik EG. Cryosurgery updated. J Am Acad Dermatol. 1994 Dec;31(6):925-44; quiz 944-6. doi: 10.1016/s0190-9622(94)70261-6. PMID 7962774
- [Background] Rodgers BM, McDonald AP, Talbert JL, Donnelly WH. Morphologic and functional effects of esophageal cryotherapy. J Thorac Cardiovasc Surg. 1979 Apr;77(4):543-9. PMID 423587
- [Background] Kantsevoy SV, Cruz-Correa MR, Vaughn CA, Jagannath SB, Pasricha PJ, Kalloo AN. Endoscopic cryotherapy for the treatment of bleeding mucosal vascular lesions of the GI tract: a pilot study. Gastrointest Endosc. 2003 Mar;57(3):403-6. doi: 10.1067/mge.2003.115. PMID 12612530
- [Background] Greenwald BD, Dumot JA, Abrams JA, Lightdale CJ, David DS, Nishioka NS, Yachimski P, Johnston MH, Shaheen NJ, Zfass AM, Smith JO, Gill KR, Burdick JS, Mallat D, Wolfsen HC. Endoscopic spray cryotherapy for esophageal cancer: safety and efficacy. Gastrointest Endosc. 2010 Apr;71(4):686-93. doi: 10.1016/j.gie.2010.01.042. PMID 20363410
- [Background] Dumot JA, Vargo JJ 2nd, Falk GW, Frey L, Lopez R, Rice TW. An open-label, prospective trial of cryospray ablation for Barrett's esophagus high-grade dysplasia and early esophageal cancer in high-risk patients. Gastrointest Endosc. 2009 Oct;70(4):635-44. doi: 10.1016/j.gie.2009.02.006. Epub 2009 Jun 25. PMID 19559428
- [Background] Finley DJ, Dycoco J, Sarkar S, Krimsky WS, Sherwood JT, Dekeratry D, Downie G, Atwood J, Fernando HC, Rusch VW. Airway spray cryotherapy: initial outcomes from a multiinstitutional registry. Ann Thorac Surg. 2012 Jul;94(1):199-203; discussion 203-4. doi: 10.1016/j.athoracsur.2012.01.112. Epub 2012 Apr 18. PMID 22516831
- [Background] Au JT, Carson J, Monette S, Finley DJ. Spray cryotherapy is effective for bronchoscopic, endoscopic and open ablation of thoracic tissues. Interact Cardiovasc Thorac Surg. 2012 Oct;15(4):580-4. doi: 10.1093/icvts/ivs192. Epub 2012 Jul 18. PMID 22811511
- [Background] Krimsky WS, Rodrigues MP, Malayaman N, Sarkar S. Spray cryotherapy for the treatment of glottic and subglottic stenosis. Laryngoscope. 2010 Mar;120(3):473-7. doi: 10.1002/lary.20794. PMID 20058314
- [Background] Fernando HC, Dekeratry D, Downie G, Finley D, Sullivan V, Sarkar S, Rivas R Jr, Santos RS. Feasibility of spray cryotherapy and balloon dilation for non-malignant strictures of the airway. Eur J Cardiothorac Surg. 2011 Nov;40(5):1177-80. doi: 10.1016/j.ejcts.2011.02.062. Epub 2011 Apr 8. PMID 21482131
- [Background] Evantash E, Hill EC, Pernoll ML. Benign disorders of the uterine cervix. Current Obstetric& Gynecologic, Diagnosis & Treatment. 9th ed. Beijing: The McGraw-Hill Companies. 2003:677-692
- [Background] Holschneider CH. Premalignant and malignant disorders of the uterine cervix. Current Diagnosis and Treatment Obstetrics and Gynecology,. 2007:833-854
- [Background] Jacob M, Broekhuizen FF, Castro W, Sellors J. Experience using cryotherapy for treatment of cervical precancerous lesions in low-resource settings. Int J Gynaecol Obstet. 2005 May;89 Suppl 2:S13-20. doi: 10.1016/j.ijgo.2005.01.026. PMID 15823262
- [Background] Stulberg DL, Crandell B, Fawcett RS. Diagnosis and treatment of basal cell and squamous cell carcinomas. Am Fam Physician. 2004 Oct 15;70(8):1481-8. PMID 15526735
- [Background] Jaros E, Priborsky J. [15 years' clinical experience in cryodestruction of malignant disorders in the anorectum]. Rozhl Chir. 1999 Sep;78(9):473-7. Czech. PMID 11077879
- [Background] Cestari A, Guazzoni G, dell'Acqua V, Nava L, Cardone G, Balconi G, Naspro R, Montorsi F, Rigatti P. Laparoscopic cryoablation of solid renal masses: intermediate term followup. J Urol. 2004 Oct;172(4 Pt 1):1267-70. doi: 10.1097/01.ju.0000140073.57974.82. PMID 15371821
- [Background] Powell T, Whelan C, Schwartz BF. Laparoscopic renal cryotherapy: biology, techniques and outcomes. Minerva Urol Nefrol. 2005 Jun;57(2):109-18. PMID 15951735
- [Background] Goldberg SR, Neifeld JP. Incidentally discovered gallbladder cancer: role of cryotherapy. J Surg Oncol. 2004 Aug 1;87(2):91-4. doi: 10.1002/jso.20075. PMID 15282703
- [Background] Dong K, Li B, Guan QL, Huang T. Analysis of multiple factors of postsurgical gastroparesis syndrome after pancreaticoduodenectomy and cryotherapy for pancreatic cancer. World J Gastroenterol. 2004 Aug 15;10(16):2434-8. doi: 10.3748/wjg.v10.i16.2434. PMID 15285038
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston MH. Cryoablation of Dysplasia in Barrett's Esophagus (BE) and Early Stage Esophageal Cancer. Gastrointestinal endoscopy. 2006;63(5):AB223
- [Background] Johnston MH. Reversal of barrett's esophagus with cryotherapy. The American journal of gastroenterology. 2003;98:S11
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Shaheen NJ, Greenwald BD, Peery AF, Dumot JA, Nishioka NS, Wolfsen HC, Burdick JS, Abrams JA, Wang KK, Mallat D, Johnston MH, Zfass AM, Smith JO, Barthel JS, Lightdale CJ. Safety and efficacy of endoscopic spray cryotherapy for Barrett's esophagus with high-grade dysplasia. Gastrointest Endosc. 2010 Apr;71(4):680-5. doi: 10.1016/j.gie.2010.01.018. PMID 20363409